CLINICAL TRIAL: NCT02986204
Title: Identification and Removal of the Non Palpable Etonogestrel Contraceptive Implant
Acronym: ENG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Angela Chen, MD, Principle Investigator, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: version 1.0 07/25/16
Record Dates: First submitted 2016-12-02; First posted 2016-12-08 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Women With an ENG Contraceptive Implant
Keywords: implant removal; Nexplanon; Implanon; contraception; ENG

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- removal of ENG implant group (Other): 20 women who have an ENG implant that is difficult to feel on exam and would like to have it removed.
  Interventions: Procedure: removal of ENG implant
- continuation of ENG implant (Other): 20 women who have are continuing to use their ENG implant.
  Interventions: Procedure: continuation of ING implant

INTERVENTIONS:
Procedure: removal of ENG implant — the researcher(s) will ask you to: Visit 1 - SCREENING VISIT
  * questions about your medical/contraception history
  * Review medical record
  * physical examination
  * urine sample for pregnancy test
  Visit 2a - Radiology
  * Have an ultrasound of your arm
  * The radiologist will mark your arm at the location of the implant.
  Visit 2b
  * ultrasound of your arm to locate the implant. This is done by feeling the area.
  * Have your ENG implant removed through a numbed small cut. The researcher will apply a pressure bandage to the site(s). This will reduce bleeding/decrease swelling.
  * Have the removal procedure video recorded.
  Visit 3 - FOLLOW UP VISIT approximately 2 weeks after Visit 2:
  * Provide a urine sample for pregnancy test
  * Have the implant removal site examined
  Arms: removal of ENG implant group
Procedure: continuation of ING implant — the researcher(s) will ask you to:
  * To answer questions about your medical and contraception history
  * Review your medical record
  * Have a physical examination by the researcher
  * Provide a urine sample for pregnancy test
  * Have an ultrasound of your arm
  Arms: continuation of ENG implant

SUMMARY:
This study will investigate in-office ultrasound localization vs localization in radiology for identification and removal of non palpable etonogestrel (ENG) contraceptive implants and aims to help establish best practices in this domain. Investigators will also create an ultrasound image gallery of palpable and non palpable as well as instructional video for non palpable ENG implant removal.

DETAILED DESCRIPTION:
This is a descriptive study to establish best practices for ENG implant localization and non-palpable ENG implant removal.

Women presenting to UCLA Obstetrics and Gynecology service for ENG non-palpable and palpable implant removal or with ENG implant in place but desiring continuation will be enrolled. Investigators aim to enroll 20 women in each group. Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria will be entered into the study.

Study duration for each participant is one visit for continuation group and two weeks for group desiring implant removal. Total study duration is expected to be 18 months.

1. For women desiring implant removal: document ENG implant using in-office imaging of ENG implant in the FP clinic with standard ob/gyn office ultrasound (abdominal 15 MHz linear probe with color doppler) and the same, using high frequency vascular probe (20+ MHz) in the radiology department.
2. Create an image gallery of office and radiology department obtained images of ENG implant localization. This will include:

   1. Ultrasound images obtained in women with palpable or non-palpable ENG implants in place at various time intervals after insertion who desire ENG implant continuation (office imaging only).
   2. Ultrasound images obtained in women seeking removal of non-palpable ENG implants, primarily referred patients who have either failed outside implant removal or have a non-palpable implant on presentation for removal.
3. Document and describe all cases of non palpable ENG implant removal with standard, in-office US versus radiology ultrasound equipment. Investigators will collect radiographic images, clinical findings, instruments used, patient characteristics (BMI, weight gain, time since of insertion), success of procedure, duration of procedure, number of attempts, final location of implant, and need for referral to general or vascular surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 - 50 years old
* English or Spanish speaking
* ENG implant in place
* Removal group

  o Women with non palpable ENG implant desiring ENG implant removal
* Continuation group o Women with palpable or non-palpable ENG implant desiring continuation

Exclusion Criteria:

* Known or suspected pregnancy
* Does not meet inclusion criteria
* Known ENG implant location outside of arm
* Current anticoagulation use (removal group only)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Creation of image gallery | 18 months
  Creating an image gallery in order to locate ENG implant using ultrasound and radiological images

SECONDARY OUTCOMES:
Creation of an instructional video and reference guide for ENG implant removal. | 18 months
  If ultrasound/radiological images are successful at locating ENG implant, this data could lead to the creation of a reference guide for other providers.

CONTACTS AND LOCATIONS:
Overall Officials: UCLA Dept. OB/GYN Div. of Family Planning, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Dept. OB/GYN, Women's Health CRU, 10833 Le Conte Ave, CHS 22-265, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mommers E, Blum GF, Gent TG, Peters KP, Sordal TS, Marintcheva-Petrova M. Nexplanon, a radiopaque etonogestrel implant in combination with a next-generation applicator: 3-year results of a noncomparative multicenter trial. Am J Obstet Gynecol. 2012 Nov;207(5):388.e1-6. doi: 10.1016/j.ajog.2012.08.002. Epub 2012 Aug 10. PMID 22939402
- [Background] Pillai M, Gazet AC, Griffiths M. Continuing need for and provision of a service for non-standard implant removal. J Fam Plann Reprod Health Care. 2014 Apr;40(2):126-32. doi: 10.1136/jfprhc-2013-100619. Epub 2013 Sep 30. PMID 24081828
- [Background] Guiahi M, Tocce K, Teal S, Green T, Rochon P. Removal of a Nexplanon implant located in the biceps muscle using a combination of ultrasound and fluoroscopy guidance. Contraception. 2014 Dec;90(6):606-8. doi: 10.1016/j.contraception.2014.06.030. Epub 2014 Jun 27. PMID 25081861
- [Background] Chen MJ, Creinin MD. Removal of a Nonpalpable Etonogestrel Implant With Preprocedure Ultrasonography and Modified Vasectomy Clamp. Obstet Gynecol. 2015 Nov;126(5):935-938. doi: 10.1097/AOG.0000000000001082. PMID 26444124
- [Background] Singh M, Mansour D, Richardson D. Location and removal of non-palpable Implanon implants with the aid of ultrasound guidance. J Fam Plann Reprod Health Care. 2006 Jul;32(3):153-6. doi: 10.1783/147118906777888549. PMID 16857066